CLINICAL TRIAL: NCT06725771
Title: Clinical Study on the Treatment of Generalized Anxiety Disorder With Chaihu Jia Longgu Muli Tang (Bupleurum Plus Dragon Bone and Oyster Shell Decoction)
Brief Title: A Non-randomized Controlled Trial Was Conducted to Observe the Improvement in the Level of HAMA in Patients With Generalized Anxiety Disorder During the 6-week Period of Oral Treatment With Chaihu Jia Longgu Muli Tang (Bupleurum Plus Dragon Bone and Oyster Shell Decoction) Combined With Sertraline.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lin Xiaoqian (Other)
Collaborators: Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Lin Xiaoqian, Jiangsu Province Hospital of TCM Affiliated Hospital of Nanjing University of Chinese Medicine, Jiangsu Province Hospital of Traditional Chinese Medicine
Organization: Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024NL-253-02
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Generalised Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Chaihu Jia Longgu Muli Tang; Sertraline; Heat-Depressed on Shao-Yang
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupleurum Plus Dragon Bone and Oyster Shell Decoction with sertraline (Experimental): observation group
  Interventions: Drug: Bupleurum Plus Dragon Bone and Oyster Shell Decoction Combined with Sertraline
- Sertraline (Active Comparator): Control group
  Interventions: Drug: Sertraline Hydrochloride Tablets

INTERVENTIONS:
Drug: Bupleurum Plus Dragon Bone and Oyster Shell Decoction Combined with Sertraline — Bupleurum Plus Dragon Bone and Oyster Shell Decoction and Sertraline are given to patients simultaneously
  Arms: Bupleurum Plus Dragon Bone and Oyster Shell Decoction with sertraline
Drug: Sertraline Hydrochloride Tablets — Sertraline are given to patients simultaneously
  Arms: Sertraline

SUMMARY:
The purpose of this study is to clinically observe the efficacy of Bupleurum Plus Dragon Bone and Oyster Shell Decoction in the treatment of Generalized Anxiety Disorder to improve the scores of HAMA

DETAILED DESCRIPTION:
Generalized Anxiety Disorder, not only results in a disturbed psychological condition, but even daily life with coworkers and family will also be disrupted. Chaihu Jia Longgu Muli Tang (Bupleurum Plus Dragon Bone and Oyster Shell Decoction), a compound Chinese herbal medicine found in "Treatise on Cold Damage", has been used for treating mental disorders with symptoms such as chest distress, irritability, being frightened, etc since the China Han dynasty. In this study, we will observe the efficacy of this formula, in order to provide an evidence-based basis for clinical observation and evaluation of Generalized Anxiety Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Meets the western medical diagnostic criteria for generalized anxiety disorder;
* The TCM diagnosis is Heat-Depressed on Shao-Yang (rè yù shǎo yáng) type;
* Hamilton Anxiety Scale (HAMA) score ≥ 7;
* Age 18-80 years old.

Exclusion Criteria:

* Allergy to Chinese Medicine formulas;
* Pregnant or breastfeeding;
* Suicidal ideation and suicide attempt;
* Substance use disorders;
* Severe cardiovascular diseases liver diseases and kidney diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Scale (HAMA) | 0, 2, 4, 6 weeks
  To evaluate participant's anxiety status

SECONDARY OUTCOMES:
Heat-Depressed on Shaoyang scale | 0, 2, 4, 6 weeks
  To evaluate participant's somatic symptoms, based on Chaihu Jia Longgu Muli Tang treatment

OTHER OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 0, 2, 4, 6 weeks
  To evaluate participant's sleep disturbances status
Hamilton Depression Scale (HAMD-24) | 0, 2, 4, 6 weeks
  To evaluate participant's depression status

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital of TCM Affiliated Hospital of Nanjing University of Chinese Medicine, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No